CLINICAL TRIAL: NCT06713759
Title: Impact of Postural Balance Changes on Low Back Pain During Pregnancy
Acronym: LBP
Status: Not yet recruiting | Type: Observational
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Nada Fawzy Ali, principle investigator: nada fawzy ali, October 6 University
Other Study IDs: P.T.REC/012/005384
Record Dates: First submitted 2024-11-28; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Pregnancy; Low Back Pain
Keywords: postural balance; low back pain; pregnacy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- primigravida women: This group will include 20 primigravida pregnant woman with low back pain. They will undergo balance and low back pain assessment (at 2 different time points: one at their second trimester (22-24) weeks and the other one in their third trimester (34th) week
- Multigravida women: This group will include 20 pregnant women with low back pain. They will undergo balance and low back pain assessment (at 2 different time points: one at their second trimester (22-24) weeks and the other one in their third trimester (34th) week

SUMMARY:
this study will be conducted to determine the impact of postural balance changes on low back pain during pregnancy

DETAILED DESCRIPTION:
Back pain is a major problem in the general population, and it is thought to be even more common in pregnant women who have given birth. It has been hypothesized that this type of pregnancy-related low back pain (LBP) may be related to changes in lumbar posture, perhaps accompanied by stretching abdominal muscles or specific hormonal effects of pregnancy .During pregnancy, many hormonal, anatomical, and musculoskeletal changes occur. These changes alter the postural balance and increase the risk of falls. Falls during pregnancy can cause maternal and foetal injuries. Moreover, the incidence of falls during pregnancy is higher compared to non-pregnant women of the same age. The risk of falls increases with the gestational age, and most falls are experienced in the third trimester. so, this study will be designed to conduct new information about the relation between postural changes and low back pain during pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in 2nd and 3rd trimesters.
* Pregnant women suffering from low back pain
* Their Age will range from 20-35 years.
* Their Body mass index (BMI) will be less than 35 kg/m2

Exclusion Criteria:

* Non pregnant women.
* Women who have any history of diseases associated with balance disorder
* Women who have any Neurological disorders.
* Women who have Lower limbs deformities
* Women who have Optical problems and disorders
* Women who have Cerebrovascular disease

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: This study will be conducted on forty pregnant women (in second and third trimesters) suffering from low back pain
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-05 (Estimated); Primary Completion 2025-02-05 (Estimated); Study Completion 2025-02-05 (Estimated)

PRIMARY OUTCOMES:
balance | up to thirty four weeks
  The Biodex Balance System SD will be used to assess balance.higher values indicate more deviations and poor balance control.
pressure pain threshold | up to thirty four weeks
  digital pressure algometer from Wagner Instruments will be used to assess pressure pain threshol.The algometer was set to measure at a rate of 100 readings per second and always displayed the highest pressure measured. The round attachment surface had a diameter of 1.12 cm. Newton (N) was set as the unit of measurement on the device. Later, it was converted to kilopascals (kPa) to enable comparability with other studies

SECONDARY OUTCOMES:
pain intensity | up to thirty four weeks
  visual analogue scale will be used to assess pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.